CLINICAL TRIAL: NCT07087470
Title: The Effect of Simulation Based Psychosocial Care Skill Development Programme on Psychosocial Care Competencies and Professional Life Quality of Oncology Nurses
Brief Title: Simulation Psychosocial Care Skills and Oncology Nursing
Acronym: SPCSAON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Collaborators: Acibadem Maslak Hospital (Other); Acıbadem Atunizade Hospital (Other); Acibadem Atakent University Hospital (Other)
Responsible Party: Principal Investigator, tülay demiray, MSc, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UU-HB-TDEMİRAY-001
Record Dates: First submitted 2025-05-01; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Simulation-based Training

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: single participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Standart psychosocial care skills training (Active Comparator): Nurses Receiving Simulation Based Training and classical psychosocial care skills training
  Interventions: Behavioral: Simulation-based education and classical education
- Group 2 (Active Comparator): only the group that will receive training in classical psychosocial care skills
  Interventions: Behavioral: classical education
- Group 3 (No Intervention): No training will be given to any group

INTERVENTIONS:
Behavioral: Simulation-based education and classical education — Simulation-based psychosocial care skills training and classical psychosocial care skills training will be prepared for oncology nurses.
  Arms: Group 1 Standart psychosocial care skills training
Behavioral: classical education — classical psychosocial care skills training will be prepared for oncology nurses.
  Arms: Group 2

SUMMARY:
The aim of this study was to reveal the effect of simulation-based experience-based psychosocial care skills development programme on psychosocial care skills competence and professional quality of life of nurses working with oncology patients.

The hypotheses of the study will be tested in accordance with the following guidelines.

Hypothesis 1 The post-training psychosocial care competency levels of the nurses who underwent simulation-based psychosocial care skills development programme (SDPBSP) are higher than the group who underwent standard psychosocial care skills training (SPBBE).

Hypothesis 2 The post-training compassion fatigue levels of the nurses who underwent the SDPBI development programme were lower than the SPBBE group.

Hypothesis 3 The post-training burnout score levels of the nurses who underwent SPBBE development programme were lower than the group who underwent standard SPBBE.

Hypothesis 4 The post-training compassion satisfaction levels of the nurses who underwent SPBBE development programme are higher than the group who underwent standard SPBBE.

Hypothesis 5

The psychosocial care competency levels of the nurses who underwent SPBBE development programme at the 1-month post-training follow-up were higher than those who did not receive SPBBE training.

Hypothesis 6 At the 1-month follow-up after the training, the compassion fatigue levels of the nurses who underwent SPBBE development programme were lower than the group who underwent SPBBE and did not receive training.

Hypothesis 7 In the 1-month follow-up after the training, the mean burnout scores of the nurses who underwent SPBBE development programme were lower than those of the group who underwent SPBBE and did not receive training.

Hypothesis 8 In the 1-month follow-up after the training, the mean compassion satisfaction scores of the nurses who underwent the SPBBE development programme were higher than the SPBBE training and non-training groups.

Hypothesis 9 After the SDPBE programme, the psychosocial skills training scores of those who received SDPBE are higher than those who did not receive training.

Hypothesis 10 At the 1-month follow-up after the SDPBE programme, the psychosocial skills training scores of those who received SDPBE were higher than those who did not receive training.

DETAILED DESCRIPTION:
The research will be applied to nurses working with oncology patients and will be randomised controlled and consist of 3 groups.

The groups will be studied as follows. Group 1: Data collection tools related to Simulation Based Psychosocial Care Skills Development Programme

* Participant Information Form
* Psychosocial Care Competence Self-Assessment Scale (PSCSAS)
* Professional Quality of Life Scale (PQLS)
* Student Satisfaction and Self-Confidence Scale in Learning
* Simulation Design Scale

Group 2: Data collection tools related to the group to be trained on Classical Psychosocial Care Skills

* Participant Information Form
* Psychosocial Care Competence Self-Assessment Scale (PSCSAS)
* Professional Quality of Life Scale (PQLS)

Group 3: Data collection tools related to the control group (group that did not receive training)

* Participant Information Form
* Psychosocial Care Competence Self-Assessment Scale (PSCSAS)
* Professional Quality of Life Scale (PQLS)

ELIGIBILITY:
Inclusion Criteria:

* 6 months or more experience of working with oncology patients
* Not having received training on psychosocial care skills after graduation
* Oncology nurses who volunteered to participate in the study

Exclusion Criteria:

* Having less than 6 months of experience working with oncology patients
* To have received training on psychosocial care skills after graduation
* Not volunteering to participate in the research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of nurses' psychosocial care competence | T1: Baseline, T2: 1. Day, T3: 1 Months post- intervention
  Psychosocial Care Competence Self-Assessment Scale (PBYÖDÖ), is a tool that assesses the psychosocial care competence of nurses working in clinics and the extent to which staff focus on the psychosocial aspects of patients while providing treatment and care. The scale, whose validity and reliability were established by Karataş (2019), consists of 18 items and 4 factors (sub-dimensions). The first factor, "Symptom Diagnosis," includes statements 1, 2, 3, 4, and 5, which are related to symptom diagnosis, for a total of 5 items. The second factor, "Use of Information," includes statements 6, 7, 8, 9, and 10, which are related to the use of information and comprise a total of 5 items. The third factor, "Intervention," includes statements 11, 12, 13, and 14, which are related to the use of information and comprise a total of 4 items. The fourth factor, "Diagnosis," includes statements 15, 16, 17, and 18, which are related to diagnosis and cover a total of 4 items. Respondents ar
Evaluation of Student Satisfaction and Self-Confidence in Learning in Simulation Applications | T1: Baseline, T2: 1 day post education, TE: 1 Months post intervention
  Student Satisfaction and Self-Confidence Scale in Learning: The psychometric measurements of the scale developed by Jeffries (2012) to assess student satisfaction and self-confidence and used in simulation-based education were conducted by Franklin et al. (2014). The Turkish validity and reliability study of the scale was conducted by Ünver et al. (2017). According to the Turkish adaptation of the scale for learning in a simulation environment, the total number of items is 12. The scale consists of two subheadings: "Satisfaction with Current Learning" and "Confidence in Learning." The "Satisfaction with Current Learning" subheading consists of five items, while the "Confidence in Learning" subheading consists of seven items. There are no negative items in the scale. A 5-point Likert scale with the following statements was used: 1) Strongly Disagree, 2) Disagree, 3) Undecided, 4) Agree, and 5) Strongly Agree. The Cronbach Alpha value for "Current Learning Satisfaction" is 0.85, and the
Assessment of nurses' professional quality of life | T1: Baseline, T2: 1 day post education, TE: 1 Months post intervention
  Professional Quality of Life Scale (PYKÖ) was developed by Stamm (2005) and consists of the subdimensions of compassion satisfaction, compassion fatigue, and burnout. The Turkish adaptation of the scale was conducted by Yeşil et al. (2010) and consists of thirty items and three subscales. Compassion satisfaction (job satisfaction) is the first of the subscales and refers to the sense of satisfaction and contentment an employee feels as a result of helping another person in need in their profession or job. Items 3, 6, 12, 16, 18, 20, 22, 24, 27, and 30 on the scale measure job satisfaction (Min 0-Max 50). A high score on this subscale indicates increased satisfaction or fulfillment as a helper. The second subscale, burnout, is a test that measures feelings of exhaustion arising from difficulties in coping with problems in work life. Items 1, 4, 8, 10, 15, 17, 19, 21, 26, and 29 on the scale measure burnout (Min 0-Max 25). A high score on this subscale indicates a high level of burnout

OTHER OUTCOMES:
Evaluation of simulation design | T1: Baseline, T2: 1 day post education, T3: 1 Months post intervention
  The scale consists of 20 items and five subscales 'Goals and Knowledge', 'Support', 'Problem Solving', 'Feedback/Guided Reflection', 'Fidelity'. 'Goals and Knowledge' subscale consists of five items, "Support" subscale consists of four items, "Problem Solving" subscale consists of five items, "Feedback/Guided Reflection" subscale consists of four items, and "Fidelity" subscale consists of two items. The scale consists of two parts. In the first part, it is measured whether the best simulation design elements are applied in the simulation application.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Tülay Demiray, Istanbul, Turkey
  - Acibadem Altunizade Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No